CLINICAL TRIAL: NCT00865202
Title: A Placebo Controlled Trial Of L-Tryptophan In Post-Operative Delirium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-0543
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Post-operative Delirium
Keywords: delirium; surgery; operation; geriatric; complication
MeSH Terms: conditions — Emergence Delirium; Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-Tryptophan (Experimental): L-tryptophan supplementation (1 gram enterally three times per day) starting post-operatively and continuing for a maximum of 9 doses or the time of discharge from ICU (whichever occurs first)
  Interventions: Drug: L-tryptophan supplementation
- Placebo (Placebo Comparator): Similar appearing placebo administered post-operatively (1 enterally three times per day) for a total of nine doses or discharge from ICU (whichever occurs first)
  Interventions: Drug: L-tryptophan supplementation; Drug: placebo

INTERVENTIONS:
Drug: L-tryptophan supplementation — L-tryptophan 1 gram enterally TID for a maximum of nine doses or to be discontinued at the time of discharge from the ICU (whichever occurs first)
  Other Names: L-tryptophan 1 gm PO TID starting the evening of surgery
Drug: placebo — Similar appearing placebo administered post-operatively (1 enterally TID) for a total of nine doses or discharge from ICU (whichever occurs first)
  Other Names: Similar appearing placebo
  Arms: Placebo

SUMMARY:
Post-operative delirium is a common and deleterious complication in elderly patients. The investigators have previously found lower levels of serum tryptophan in post-operative elderly patients who developed delirium in comparison to post-operative elderly patients who did not develop delirium. The investigators hypothesize that post-operative supplementation of L-tryptophan will reduce the duration and incidence of post-operative delirium. This study is a double-blinded placebo controlled trial of L-tryptophan supplementation in post-operative ICU patients 60 years and older. The primary outcome measure is the comparison of duration of post-operative delirium in subjects who receive L-tryptophan supplementation versus a similar appearing control.

DETAILED DESCRIPTION:
The sudy will compare rates and duration of postoperative delirium in groups that receive L-tryptophan supplementation compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Included subjects will be 60 years and older undergoing an operation with a planned ICU admission post-operatively.

Exclusion Criteria:

* Medications that, when combined with tryptophan, increase the risk of serotonin syndrome. The classes of medications include:

  * monoamine oxidase inhibitors
  * selective serotonin reuptake inhibitors
  * serotonin-norepinephrine reuptake inhibitors
  * triptans
  * opioids
  * central nervous system stimulants
  * bupropion
  * St. John's Wort
* Patients who undergo an operation on their brain.
* Factors which prevent delirium assessment with the CAM-ICU: vision impairment or non-fluent English speakers.
* A lowered seizure threshold including:

  * history of seizure disorder
  * alcohol abuse defined by a high AUDIT score (>8 females and >13 males)
  * benzodiazepine or barbiturate abuse within three months of the study
  * OR a positive urine toxicology screen for alcohol, benzodiazepines or barbiturates.
* Significant liver disease (Child's class B or greater) or significant renal disease (Creatinine ≥2.0).
* History of Huntington's or Addison's disease. (As requested by the FDA)
* History of bipolar disorder or a psychotic disorder (such as a psychotic major depression, schizophrenia, schizoaffective disorder, or psychosis in Alzheimer's disease or other dementia). (As requested by the FDA)
* Women who are not post-menopausal. (As requested by the FDA)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Robinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Denver Veterans Affairs Medical Center, Denver, Colorado, United States

REFERENCES:
- [Background] Robinson TN, Raeburn CD, Angles EM, Moss M. Low tryptophan levels are associated with postoperative delirium in the elderly. Am J Surg. 2008 Nov;196(5):670-4. doi: 10.1016/j.amjsurg.2008.07.007. Epub 2008 Sep 11. PMID 18789427
- [Background] Robinson TN, Raeburn CD, Tran ZV, Angles EM, Brenner LA, Moss M. Postoperative delirium in the elderly: risk factors and outcomes. Ann Surg. 2009 Jan;249(1):173-8. doi: 10.1097/SLA.0b013e31818e4776. PMID 19106695

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Drug: L-tryptophan 1 gm enterally TID starting the evening of the operation
- Placebo: Similar appearing placebo
Period: Overall Study
Arm/Group | Study Drug | Placebo
Started | 152 | 149
Completed | 152 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 301 total study participants
Groups:
- L-tryptophan: L-tryptophan 1 gm enterally TID starting the evening of the operation
- Total: Total of all reporting groups
Arm/Group | L-tryptophan | Placebo | Total
Number analyzed (Participants) | 152 | 149 | 301
Age, Continuous [Mean (Standard Deviation); unit: years]
  Overall Study | 69 (7) | 69 (8) | 69 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 148 | 147 | 295
Region of Enrollment [Number; unit: participants]
  United States | 152 | 149 | 301

OUTCOME MEASURES:

1. Primary Outcome: Duration of Post-operative Delirium
Time Frame: post-operatively daily in ICU until discharged from ICU
Measure: Mean (Standard Deviation); unit: days
Groups:
- Study Drug: L-tryptophan 1 gm PO TID starting the evening of surgery
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 152 | 149
days | 3.3 (1.7) | 3.1 (1.9)

2. Secondary Outcome: Incidence of Post-operative Delirium
Description: The incidence and/or duration of excitatory (hyperactive and mixed) post-operative delirium, diagnosed by the Confusion Assessment Method-ICU (CAM-ICU) with the Richmond Agitation Sedation Score (RASS), will be reduced with enteral L-tryptophan supplementation (1 gm TID for the first 3 post-op days), compared to placebo, in older patients (≥ 60 years) undergoing operations requiring ICU admission.
  The incidence and/or duration of all types of post-operative delirium, diagnosed by the CAM-ICU with the RASS, will be reduced with enteral L-tryptophan supplementation (1 gm TID for the first 3 post-op days), compared to placebo, in older patients (≥ 60 years) undergoing operations requiring ICU admission.
Time Frame: post-operatively daily in ICU until discharged from ICU
Measure: Number; unit: percentage of patient escitatorydelirium
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 152 | 149
percentage of patient escitatorydelirium | 17 | 9

3. Secondary Outcome: Level of Post-operative Serum Tryptophan
Time Frame: post-operative day number two blood draw
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 152 | 149
umol/L | 65 (26) | 41 (15)

4. Secondary Outcome: Level of Post-operative Melatonin
Time Frame: Blood draw on post-operative day number two
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 152 | 149
pg/mL | 20 (31) | 19 (41)

5. Secondary Outcome: Length of Post-operative ICU and Hospital Stay
Time Frame: length of post-op hospital stay
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Study Drug | Placebo
Number analyzed (Participants) | 152 | 149
days | 10 (8.4) | 9.7 (8.7)

ADVERSE EVENTS:
Time Frame: Postoperative Nausea
Description: Postoperative Nausea
Arm/Group | Study Drug | Placebo
Serious Adverse Events (participants affected / at risk) | 0/152 | 0/149
Other Adverse Events (participants affected / at risk) | 0/152 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The manuscript has been accepted by the Journal of the American Geriatrics Society for publication.